CLINICAL TRIAL: NCT03656497
Title: Classical Trigeminal Neuralgia and Sodium Channel Mutations
Status: Completed | Type: Observational
Sponsor: Danish Headache Center (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Tone Heinskou, MD, PhD student, Danish Headache Center
Other Study IDs: H-15010165
Record Dates: First submitted 2018-08-29; First posted 2018-09-04 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Trigeminal Neuralgia
Keywords: genetic mutations, voltage gated sodium channels, phenotype,
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — full blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — No intervention is conducted as the study aim is to explore the link between pheno- and genetype of trigeminal neuralgia

SUMMARY:
The most common cause of trigeminal neuralgia is considered to be a neurovascular contact. However, this etiological factor only seem to be present in half of the patient group. Thus the etiology of the other half is unknown.

Gain-of function genetic mutations in voltage gated sodium channels have been hypothesized as playing a role in the etiology of trigeminal neuralgia but it has yet to be confirmed. In recent years gain-of-function mutations have been identified as a causative factor in other pain-diseases presenting with trigeminal neuralgia phenotypic similarities.

DETAILED DESCRIPTION:
The aim of this study was to indentify VGSC gene mutations, specifically SCN9A, SCN10A and SCN11A genes, in a group of well characterized trigeminal neuralgia patients.

Setting: The study will be conducted at The Danish Headache Center, Rigshospitalet - Glostrup, Denmark (inclusion of patients and written Informed Consent, patient interview, phenotyping/diagnosis, neurological examination, blood sample.

Departments of Neurology and Clinical Genomics of the Maastricht University Medical Center, Maastricht, the Netherlands: Targeted NG Sanger Sequencing

ELIGIBILITY:
3.1. Inclusion Criteria

Subjects of both sexes with TN must meet the following inclusion criteria to be eligible for participation:

1. Patients must be able to give Signed Informed Consent prior to study entry
2. Patients fulfilling of the ICHD-3 beta diagnostic criteria for classical TN.1
3. Age 18 years or older.
4. Age at debut < 42 years and/or confirmed first-line relative with TN.
5. Respond to sodium channel blockers with a 50% reduction of pain intensity evaluated by both the patient and the examining physician using the visual analog scale (VAS).

3.2. Exclusion Criteria

Subjects will be excluded if one of the following exclusion criteria is met:

1. Psychiatric or mental illness of physical condition that might interfere with the ability of the patients to fill in the Informed Consent and questionnaires.
2. History of herpes zoster in the distribution of the trigeminal nerve ipsilateral to pain, multiple sclerosis or a space-occupying lesion.
3. History indicative of painful posttraumatic trigeminal neuropathy such as previous trauma, surgery or radiation to the trigeminal nerve ipsilateral to pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from trigeminal neuralgia and has an onset of disease before the age of 42 and/or first-line relative with TN.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Exploratory study of association between phenotype and genotype of trigeminal neuralgia | 1 day
  To identify genetic mutations, via Sanger Next Generation Sequencing, in either NaV 1.7, NaV1.8 or NaV1.9 encoding genes and link the findings to the phenotype of trigeminal neurlagia patients with a high genetic load.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bendtsen, ass. prof., Study Chair — Danish Headache Center

IPD SHARING:
Plan to Share IPD: Undecided